CLINICAL TRIAL: NCT01527344
Title: Assessment of Cardiac Allograft Vasculopathy With Optical Coherence Tomography as Compared to Intravascular Ultrasound-Virtual Histology
Brief Title: Assessment of Cardiac Allograft Vasculopathy With Optical Coherence Tomography
Acronym: CAV-OCT-IVUS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Amir Lerman, MD, Mayo Clinic
Other Study IDs: 11-003775
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: OCT; IVUS; CAV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiac allograft vasculopathy (CAV) is a progressive disease of the coronary arteries in transplanted hearts which is a significant cause of morbidity and mortality. The broad objective of this research study is to advance our ability to diagnose as early as possible the presence of CAV and to non-invasively predict those patients at increased risk of CAV with novel techniques. Optical coherence tomography (OCT) is a novel intracoronary imaging technique using an optical analog of ultrasound with a resolution 10 times greater resolution than intravascular ultrasound (IVUS). Endothelial progenitor cells (EPCs) in peripheral blood have been shown to play a role in the pathogenesis of atherosclerosis and peripheral arterial tonometry is a clinical tool used to predict endothelial dysfunction (a precursor of atherosclerosis) which has been validated in non-transplant patients. Patients scheduled for routine cardiac catheterization with IVUS at the Mayo Clinic Rochester, Minnesota (MN) that reach inclusion and exclusion criteria for the study will be approached on the day to get informed consent to perform OCT, blood sampling and peripheral endothelial function testing. The investigators aim to 1) compare the frequency and plaque type of CAV as defined with OCT versus IVUS-Virtual Histology (IVUS-VH), 2) predict the presence and severity of CAV with absolute counts of EPCs and 3) with peripheral endothelial function scores.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older
* patients with cardiac transplant undergoing routine CAV surveillance

Exclusion Criteria:

* patients < 18 years old
* patients with acute rejection
* patients with active infection
* patients with chronic renal insufficiency with a glomerular filtration rate (GFR) < 30ml/min
* patients not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplant Patients
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Characterize CAV in-vivo with OCT | 1 year

SECONDARY OUTCOMES:
Compare the frequency and plaque type of CAV as defined with OCT versus IVUS-VH | 1 year
Predict the presence and severity of CAV with absolute counts of EPCs. | 1 year
Predict the presence and severity of CAV with peripheral endothelial function scores | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Cardiovascular Diseases, Professor of Medicine, Mayo Clinic Rochester
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States